CLINICAL TRIAL: NCT03134274
Title: Healthy.io Urine Dipstick Home Testing: a Pilot Study Among Pregnant Women
Brief Title: Study Assessing the Usability and Patient Satisfaction With Digital Urinalysis in the Context of Routine Pre-natal Care.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Healthy.io Ltd. (Industry)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HealthyioJH
Record Dates: First submitted 2017-04-24; First posted 2017-04-28 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Pregnancy

STUDY DESIGN:
Intervention Model Description: Assess usability and preference of digital home urine testing with pregnant women. 300 pregnant women will be given a test kit and smartphone application during a clinic visit. Participants are instructed to conduct the test the next day. After conducting the urine test home participants fill out a survey assessing the satisfaction with digital home urine testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Pregnant women (Experimental): Pregnant women above the age of 18 years, undergoing routine pre-natal care, who own and are familiar with use of a smartphone receive a Dip HBDA kit for home use.
  Interventions: Device: Dip HBDA

INTERVENTIONS:
Device: Dip HBDA — Participant receive Dip HBDA semiquantitative urinalyiss kit to be used at home one day after routine prenatal consultation. Dip HBDA consists of a testing kit containing calibration color board, 10 parameter urine dipstick and a urine cup as well as a smartphone application. Application guides participant through the test flow. Dipstick is immersed in urine cup, placed on color board and scanned with smartphone.

SUMMARY:
The study is a home-based, usability study assessing the use of the Dip Home-Based Dipstick Analyzer (HBDA) in the context of prenatal care.

DETAILED DESCRIPTION:
300 pregnant women receive home testing kit and smartphone application (Dip HBDA) during regular prenatal visit. They are instructed to conduct a urine test (regular 10 parameter dipstick included in kit) at home using the Dip HBDA. After conducting the urine test, participants are to fill out a short questionnaire regarding ease of use, preference of testing and any problems encountered.

This study only assesses usability and questionnaire outcomes. The results of the test (indications on dipstick) are not subject to the study.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Own and are familiar with use of a smartphone

Exclusion Criteria:

* They do not have use of both hands.
* Are visually impaired (cannot read user manual)
* Have dementia or mental disorder.
* Are not able to fill urine receptacle.
* Are not willing to adhere to study procedures.
* Do not own or are not familiar with the use of a smartphone.
* Have no access to a wifi / or cellular data connection at their home.
* Have impaired vision that prevents them from reading instructions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-05-07 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Ease of use and preference questionnaire | 2-3 months
  Questionnaire contains:
  * Ease of use among pregnant women (Ease of use ranking 1-5 measured)
  * Problems encountered while doing the test
  * Likelihood that digital home urine testing would be recommended (Net Promoter Score)
  * Preference of home testing compared to traditional testing (Prefer home testing, no preference, prefer traditional testing)

SECONDARY OUTCOMES:
Usability of Dip HBDA | 2-3 months
  Success rate in conducting the test at home (i.e. successfully completed/total participants)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Burke, MD, Principal Investigator — Johns Hopkins Medical
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No